CLINICAL TRIAL: NCT01840930
Title: Longitudinal Study of a Children Population With Bilateral Severe Cerebral Palsy: Incidence and Evolution of Orthopaedic Complications and Pain Related With These Complications.
Brief Title: Cohort of Children With Severe Cerebral Palsy
Acronym: CPCohort
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: D50687
Record Dates: First submitted 2013-04-05; First posted 2013-04-26 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Orthopedic Complications in Cerebral Palsy
Keywords: Cohort; Cerebral Palsy; Children; Pain; Orthopedic complications; Epidemiology
MeSH Terms: conditions — Cerebral Palsy; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
" Cohort CP " is a multicentre cohort study, initiated by the Hospices Civils de Lyon in September 2009. Population targeted are children with bilateral cerebral palsy, level GMFCS IV or V, aged from 2 to 10 years at inclusion. They are followed-up during 10 years, at the rhythm of 1 visit per year. At each visit are collected clinical, orthopaedic, radiological and environmental data.

The primary objective is to establish the incidence of orthopaedic complications (scoliosis and hip joint) depending on patients' age.

Secondary objectives are to describe the sequences over time of these complications and the related pain, to explore the impact of nutrition, surgery, asymmetric postures and environmental factors, and to describe the medical and rehabilitative follow-up of these patients.

385 patients are expected by the end of 2020. We expect of this long-term follow-up to gain tools that permit to improve patient's care and patient's quality of life, by putting in place preventing actions and adapted treatments related to their own pathologies.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 2 to 10 years at inclusion,
* with bilateral cerebral palsy,
* Grade IV or V of the GMFCS.
* Affiliated with the French healthcare system.
* Oral consent of the parents obtained.

Exclusion Criteria:

- Progressive pathology.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged from 2 to 10 years, with severe cerebral palsy: who do not acquire the ability to walk.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Estimated)
Dates: Start 2009-09 (Actual); Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change of hip migration (%) and/or scoliosis (Cobb angle) during the 10 years of patients' follow-up. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Hip migration is measured in percentage (Rimers method), and scoliosis is measured in degrees (Cobb angle).
  For the first visit (A00= inclusion), if hip migration measured on the last radiography is ≥ 20%, it is asked to trace the history of the migration with measurements of previous patient's radiographies. For this first visit, if the Cobb angle on the last radiography is ≥ 20°, it is also asked to trace history of scoliosis with previous radiographies.
  For the following visits (A01 to A10), only the last radiography is required for each year.

SECONDARY OUTCOMES:
Impact of nutrition on the occurrence of orthopedic complications and related pain. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Occurrence of hip migration or scoliosis correlated with annual measurement of nutritional state. Nutritional state is measured by weight, size, skinfold, and description of alimentation mode.
Impact of surgical treatment of hip luxation on pain. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Subjects split into 2 groups: pain / without pain; comparison of percentages of children operated into each group.
Impact of asymmetric postures on the occurrence of orthopedic complications and related pain. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Frequency of windswept attitude function of type of bearings and postures.
Relationship between neurological asymmetry and windswept and/or hip joint. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Frequency of neurological asymmetry function of windswept laterality and/or hip joint.
Relationship between environmental factors and orthopedic complications, pain, and nutrition. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Correlation between patient's environment, hip migration and scoliosis, pain and nutrition.
Description of the rehabilitative and medical follow-up in the studied population. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Recording of the main steps of medical and rehabilitative care received by each patient.
Description of the sequences over time of orthopedic complications and the related pain. | Day 0, year 1, year 2, year 3, year 4, year 5, year 6, year 7, year 8, year 9, year 10
  Pattern of individual evolution of pain function of age, and quantification of orthopedic surgery impact on pain evolution.
  Pain is measured with the DESS scale (Douleur Enfant San Salvadour) for children with no oral language, or with the VAS (Visual Analogue Scale) for children who have an oral language. In addition, the location, the frequency and the length of time of the related pain are recorded on the Case Report Form.

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle POIROT, PhD, Principal Investigator — Hospices Civils de Lyon - Hôpital Femme Mère Enfant
Locations (1):
- Hospices Civils de Lyon - Hôpital Femme Mère Enfant, Bron, France